CLINICAL TRIAL: NCT03442803
Title: Propofol Target-controlled Infusion Versus Usual Care for the Sedation of Adult Patients With Acute Shoulder Dislocation in the Emergency Department
Brief Title: Propofol Target-Controlled Infusion in Emergency Department Sedation
Acronym: ProTEDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GN16AE183
Record Dates: First submitted 2018-02-12; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Shoulder Dislocation
Keywords: sedation; Emergency Department; Target Controlled infusion; propofol
MeSH Terms: conditions — Shoulder Dislocation; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Propofol TCI (Experimental): Delivery of Propofol via a Target-controlled infusion pump for procedural sedation.
  Interventions: Device: Target-Controlled Infusion

INTERVENTIONS:
Device: Target-Controlled Infusion — Propofol Target-Controlled Infusion

SUMMARY:
There exists continued controversy over the use of propofol in Emergency Department procedural sedation, this is despite its widespread existence in clinical practice for at least a decade. These concerns are not limited to the ED setting and are primarily related to the pharmacological properties of the drug itself and its potential for harm. The bolus administration of propofol, aimed at a target of sedation, offers several advantages over more traditional agents, yet these advantages are also its limitations. The use of a target-controlled infusion may provide the sedationist with greater control over the pharmacokinetics of propofol and thus reduce the rate of adverse incidents.

This feasibility study aims to use a pragmatic design to test the safety and efficacy of propofol TCI whilst assessing the practicalities of it's use in the ED. If it proves to be feasible then the researchers plan to proceed to a multi centre pilot study to gather information to adequately power a larger randomised multi centre trial.

DETAILED DESCRIPTION:
Procedural sedation and analgesia (PSA) has long been a core skill of the Emergency Physician, although over the last decade, developments in patient monitoring and the use of newer sedative and analgesic agents have served to improve both safety and efficacy. Despite these advances and their consolidation into well-designed guidelines concern regarding the safety of ED PSA persists.

More specifically, concerns have been raised regarding the use of propofol, an ultra-short acting anaesthetic agent. The practice of using sub-anaesthetic doses of propofol to achieve sedation in ED PSA originated around the turn of the millennium and has since become the most common choice of sedative in the ED. Propofol offers a number of advantages as a sedative agent, including; a short onset and recovery time, amnesiac properties and good efficacy. The cost of these properties is in part, a narrow therapeutic range.

When given as a bolus, propofol will induce a spectrum of states up to and including general anaesthesia, dependent on the dosage. The correlation between dose and effect varies based on several patient factors. Whilst targeting a state of sedation it is possible for the operator to 'overshoot' moving rapidly from Conscious Sedation to Deep Sedation to General Anaesthesia. The inadvertent induction of general anesthesia may result in unanticipated complication.

The principle complications associated with accidental over-sedation or general anesthesia relate to the patency of the patient's airway. The reported frequency of airway complications during ED PSA with propofol range from 5.0% to 9.4%7, this includes a rate of supplemental ventilation of between 3.0% and 9.4%, with oxygen desaturation occurring in between 5% and 7% of cases12. In addition, the bolus administration of propofol may result in transient hypotension. Despite being a relatively short lived effect, this may be pronounced in those with intravascular volume depletion or in the elderly, and in some may be profound, with one series demonstrating that 3.5% of those undergoing PSA with propofol experience ≥ 20% falls in blood pressure. At first inspection the reported rate of complication may appear low, and has by some been interpreted as evidence of the relative safety of ED PSA, however alternative views have been expressed in the context of much lower rates of adverse events seen in elective painful procedures requiring conscious sedation. This is compounded by the non-standard way in which adverse events have been reported across studies.

A potential solution to the adverse events experienced with the bolus administration of propofol is the use of a target-controlled infusion (TCI). This method is widely used in anaesthetic practice and whilst the PK remains the same irrespective of if you give a bolus or infusion of propofol, TCI allows the titration in perhaps a more controlled manner.

The aim when administering propofol, as with any drug, is to induce a desired clinical effect, in this context a level of sedation. As previously alluded to, when administering propofol in a bolus fashion or as a fixed rate infusion, without regard to those factors which cause biologic variability (e.g. age, gender, weight), it is difficult to accurately and consistently predict clinical effect. The development, in the early 1990's, of computer assisted infusion devices, for the first time, allowed the clinician to target a plasma concentration, with the pump automatically altering the rate of infusion based on a pre-programmed pharmacokinetic model. These target-controlled infusion (TCI) devices have undergone significant development and are now in widespread clinical use. Their operation uses a mathematical mode that reflects a theoretical 'three-compartment' model that may comprise the central compartment (plasma), and two peripheral compartments (highly perfused tissue e.g. brain and poorly perfused tissue e.g. adipose). In a state of equilibrium, propofol will diffuse between compartments at a constant rate. These rate constants have been used in pharmacokinetic models to mathematically predict the plasma concentration and latterly the effect site concentration, in this case that in the brain.

In practical terms, TCI allows the operator to more accurately target a specific clinical effect. When propofol is administered as a bolus, the operator is likely to either under-dose, delivering an insufficient effect site concentration, or over-dose, exceeding the desired effect site concentration. TCI allows the operator to titrate to effect and then to maintain a steady state, potentially eliminating the risk of 'over shooting' and reducing the rate of adverse events. TCI is not without limitation. PK models are an estimate as they have been derived from a healthy population but any inherent inaccuracy is consistent in different populations and accounted for by careful titration.

The use of propofol TCI has been studied in a number of settings, including gastrointestinal endoscopy, dental surgery, oocyte retrieval and bronchoscopy. To our knowledge propofol TCI in sedation has not been studied in an ED setting. Trials have demonstrated a good safety profile for propofol TCI, with at least one large randomised-controlled trial in an endoscopy setting, showing a reduction in both respiratory and cardiovascular adverse events in comparison to the bolus administration of propofol. Unfortunately, trials to date have suffered from a high degree of heterogeneity, leading the Cochrane review, on the subject of propofol TCI versus manually controlled infusion in both general anaesthesia and sedation, to conclude that there was insufficient evidence to make firm recommendations regarding its use in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* Clinical and/or radiological evidence of acute anterior shoulder dislocation
* ASA I or II
* Fasted ≥ 90mins2,3,27,28
* Weight ≥50kg

Exclusion Criteria:

* Inability to provide or refusal of informed consent
* Previous attempt at reduction during the same presentation
* Previously enrolled in the study
* Clinical and/or radiological evidence of acute posterior shoulder dislocation
* Clinical and/or radiological evidence of concomitant ipsilateral upper limb fracture (with the exception of an isolated avulsion fracture of the greater tuberosity or a fracture of the glenoid labrum)
* Concomitant multi-system injury
* History of difficult intubation/airway surgery
* ASA grade III, IV or V
* Haemodynamic instability
* Pregnancy
* Contraindication to sedation
* Allergy to study drugs or eggs
* Clinician decision
* Morphine administration within the preceding 20minutes prior to starting TCI (can be included if >20minutes)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | Patient satisfaction will be assessed when patient is fully awake, this will be recorded on one single occasion, on average 30minutes after the procedure.
  Patient satisfaction score using a VAS with the question, "How satisfied were you with the procedure? Please mark on the line below with a vertical mark." The scale ranges from not satisfied to very satisfied.

SECONDARY OUTCOMES:
Nursing Opinion of the Patient Experience | Immediately after procedure
  Nursing opinion of the Patient experience using a VAS with the question "How would you rate the patient's experience of the procedure whilst sedated? Please mark on the line below with a vertical mark." The scale ranges from poor experience to excellent experience.
Incidence and severity of adverse events per World Society of Intravenous Anaesthesia adverse event reporting tool | Duration of sedation, on average 40 minutes
  A standardised adverse event reporting tool that categories the outcome and severity of adverse events. Outcomes can either be minimal risk outcome, moderate risk outcome, sentinel outcome or other. The severity will either be sentinel adverse event, moderate risk adverse event, minor risk adverse event or minimal risk adverse event.
Time from commencement of sedation to fit for discharge as per Royal College of Emergency Medicine guidelines outlining fit for discharge. | End of the patient's Emergency Department attendance post procedure and prior to discharge, on average 3 hours.
  Time in minutes taken for the patient to be fit for discharge after commencement of sedation, completion of procedure and cessation of sedation.
  A patient is deemed fit for discharge when they have satisfied the following criteria as defined by the Royal College of Emergency Medicine:
  * Patient returned to their baseline level of consciousness
  * Vital signs are within normal limits for that patient.
  * Respiratory status is not compromised.
  * Pain and discomfort have been addressed.
  * Patient returned to their baseline level of consciousness
  * Vital signs are within normal limits for that patient.
  * Respiratory status is not compromised.
  * Pain and discomfort have been addressed.
% of patients recruited vs % of patients approached | At the point in their attendance when approached for consent to be recruited, on average 30 minutes into their attendance.
  % of patients recruited vs % of patients approached

CONTACTS AND LOCATIONS:
Overall Officials: Fiona M Burton, MBChB, FRECM, Principal Investigator — Hairmyres Hospital
Locations (4):
- United Kingdom (4):
  - Glasgow Royal Infirmary, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - Hairmyres Hospital, Glasgow
  - Royal Alexandra Hospital, Paisley

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burton FM, Lowe DJ, Millar J, Corfield AR, Watson MJ, Sim MAB. Propofol Target-Controlled Infusion in Emergency Department Sedation (ProTEDS): a multicentre, single-arm feasibility study. Emerg Med J. 2021 Mar;38(3):205-210. doi: 10.1136/emermed-2020-209686. Epub 2020 Dec 9. PMID 33298604
- [Derived] Burton FM, Lowe DJ, Millar J, Corfield AR, Sim MAB. A study protocol for a feasibility study: Propofol Target-Controlled Infusion in Emergency Department Sedation (ProTEDS)-a multi-centre feasibility study protocol. Pilot Feasibility Stud. 2019 Feb 18;5:27. doi: 10.1186/s40814-019-0412-y. eCollection 2019. PMID 30820338